CLINICAL TRIAL: NCT02027922
Title: Randomized Clinical Trial Comparing the Clinical Effectiveness of Various Professionally Applied Fluoride Prophylaxes in Deciduous Teeth in Groups at High Risk
Brief Title: Clinical Effectiveness of Various Professionally Applied Fluoride Prophylaxes in Groups at High Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Anna Turska Szybka, Prof Ass., Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clinical effectiveness of FV
Record Dates: First submitted 2013-11-14; First posted 2014-01-06 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: White Spot Lesion; Caries
Keywords: white spot lesion; caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluoride varnish Fluor Protector S (Experimental): Fluoride varnish Fluor Protector S (Ivoclar Vivadent) with 1.5% ammonium fluoride was not scored. The emergence of a new varnish implies the necessity to compare the effectiveness of both agents in preventing caries in deciduous teeth. All of the elements of a clinical trial and the varnish applications will be performed four times at three-month intervals: examination - 0 (initial score), follow-ups to the initial examination and intervention: 1 - after 3 months, 2 - after 6 months, 3 - after 9 months. Changes in OHI-S, spot carious lesion discovered at the initial assessment as invisible, visible and inactive, active, cavities), dmft and dmfs, and their components will be scored at follow-up examinations.
  Interventions: Other: Fluor Protector S
- Duraphat (Active Comparator): 5% Sodium fluoride varnish Duraphat Colgate implies the necessity to compare the effectiveness with Fluor Protector S in preventing caries in deciduous teeth. All of the elements of a clinical trial and the varnish applications will be performed four times at three-month intervals: examination - 0 (initial score), follow-ups to the initial examination and intervention: 1 - after 3 months, 2 - after 6 months, 3 - after 9 months. Changes in OHI-S, spot carious lesion discovered at the initial assessment as invisible, visible and inactive, active, cavities), dmft and dmfs, and their components will be scored at follow-up examinations.
  Interventions: Other: Fluor Protector S
- an oral hygiene tutorial (No Intervention): an oral hygiene tutorial

INTERVENTIONS:
Other: Fluor Protector S — Fluor Protector S intervention group A (25 ml) Duraphat group B (25ml)
  Other Names: Duraphat Colgate
  Arms: Duraphat; Fluoride varnish Fluor Protector S

SUMMARY:
The study is to compare the prophylactic and therapeutic clinical effectiveness of two fluoride varnishes in children at high caries risk.

It was hypothesized, the use of Fluor Protector S (I) fluoride varnish in children with deciduous teeth at high risk of caries (P) reduces caries and the activity/remineralisation of carious enamel spots (transformation of White Spot Lesion into D (decay)) (O), similarly to what occurs after the use of Duraphat varnish (C).

DETAILED DESCRIPTION:
The study is to compare the prophylactic and therapeutic clinical effectiveness of two fluoride varnishes in children at high caries risk.

It was hypothesized, the use of Fluor Protector S (I) fluoride varnish in children with deciduous teeth at high risk of caries (P) reduces caries and the activity/remineralisation of carious enamel spots (transformation of White Spot Lesion into D (decay)) (O), similarly to what occurs after the use of Duraphat varnish (C).

The question set bases on a Caries Assessment by Risk Management system basing on the occurrence of major caries causative agents (biological and medical), and also of the protective/preventive ones. Questions related to the social and economical status will be left out because of the difficulty of getting them answered honestly. Teeth will be scored according to International Caries Detection System II classification, and oral hygiene according to the Greene and Vermillion simplified Oral Hygiene Index (OHI-S) (1964). Children and their parents/guardians will receive hygienic, dietary and prophylactic guidelines.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy children aged 3-5 years
* high risk of caries
* parent/legal guardian consent for participation in research study

Exclusion Criteria:

* chronic diseases or medication in medical history
* planned change of residence within a year
* aged <3, >5 years

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
the number of caries and white spot lesions in teeth treated with fluoride varnishes comparing to the control group. | 12 months
  The primary outcome were caries prevalence and increment.The primary endpoint for each individual child is whether or not there has been any occurrence of new caries lesions over the 1 year period, as measured by any increase in d3mft at 1 years of follow up compared to the d3mft at baseline (d3mft is dental decay as measured by the dmft scale in the dentine)

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Olczak-Kowalczyk, Professor, Principal Investigator — Medical University of Warsaw
Locations (1):
- Warsaw, Poland

REFERENCES:
- [Derived] Turska-Szybka A, Gozdowski D, Twetman S, Olczak-Kowalczyk D. Clinical Effect of Two Fluoride Varnishes in Caries-Active Preschool Children: A Randomized Controlled Trial. Caries Res. 2021;55(2):137-143. doi: 10.1159/000514168. Epub 2021 Mar 11. PMID 33706305